CLINICAL TRIAL: NCT05931406
Title: Effects of a Sedentary Behaviors at Work on Health in Emergency Medical Dispatchers and CODIS Operators
Brief Title: Effects of a Sedentary Behaviors at Work on Health in Emergency Medical Dispatchers and CODIS Operators (SECODIS)
Acronym: SECODIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2022 DUTHEIL; 2022-A02730-43 (Other: ANSM)
Record Dates: First submitted 2023-06-09; First posted 2023-07-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Sedentary Behavior; Occupational Stress
MeSH Terms: conditions — Sedentary Behavior; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency medical dispatchers (Experimental)
  Interventions: Behavioral: Control; Behavioral: Sit-and-stand desk; Behavioral: Cycloergometer
- Firefighter (Experimental)
  Interventions: Behavioral: Control; Behavioral: Sit-and-stand desk; Behavioral: Cycloergometer

INTERVENTIONS:
Behavioral: Control — A normal working day from of 12h
Behavioral: Sit-and-stand desk — a working day during which the participants have to get up at least 5 min/hour
Behavioral: Cycloergometer — a working day during which they can use a cycloergometer installed under the desk

SUMMARY:
The purpose of the study is to study changes in sedentary behavior following a behavioral intervention (sit-and-stand desk, and cycloergometer)

DETAILED DESCRIPTION:
Each emergency medical services dispatcher and each firefighter participates in the study for three days. A normal working day from of 12h is compared to: (i) a working day during which the participants have to get up at least 5 min/hour (sit-and-stand desk), (ii) a working day during which they can use a cycloergometer installed under the desk. Conditions will be random using Latin Square design with stratification between sequences cross-over design on occupation (EMD vs. firefighters).

The heart rate variability (measured using Zephyr®), the electrodermal activity (Empatica® E4), the level of physical activity (Actigraph®) as well as the blood sugar (Freestyle®) will be measured continuously during the 12 hours of work and the night after except for Actigraph® and Freestyle® device that will be let one week. Blood and saliva samples will be collected on each working day, at the beginning and end of the day i.e. two measures for blood samples, and every three hours i.e. 5 measures for saliva sampling. Participants will have to complete a detailed questionnaire to identify the particular events (vital emergencies, etc.) that may influence the parameters measured.

Participants will be asked to answer a general questionnaire once at the start of the study that will cover different aspects:

* Sociodemographic,
* Visual analogue scale (VAS) related to psychosocial factors : stress at home, burnout / burnout, decision latitude / autonomy at work, psychological demands at work (workload), support from the hierarchy, support from co-workers, family support, job satisfaction with regard to effort, commitment to work, addiction to work, quality of life, need for psychological support,
* Eating habits.

They will then have to answer a short questionnaire at the beginning and at the end of each measurement day. It will cover different aspects:

* Four VAS (stress level, fatigue, anxiety, mood),
* Physical activity and sedentary lifestyle (number of hours of physical activity and sitting during the last 24 hours),
* Daily consumption (tobacco, alcohol, cannabis, coffee, tea).

ELIGIBILITY:
Inclusion Criteria:

* Emergency medical dispatchers or firefighters from the departmental fire and rescue operational center (CODIS).
* Person able to give an informed consent to participate in research
* Affiliated with a Social Security scheme.
* Being able to use the sit-stand desk and the cycle ergometer

Exclusion Criteria:

* Non-affiliated to a health insurance,
* Protected persons (minors, pregnant women, breastfeeding women, guardianship, curatorship, deprived of freedoms, safeguard of justice),
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sedentary behavior | 12 hours of work corresponding to the control condition
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes per day standing/active.
Sedentary behavior | 12 hours of work corresponding to the sit-and-stand desk condition
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes per day standing/active.
Sedentary behavior | 12 hours of work corresponding to the cycloergometer condition
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes per day standing/active.

SECONDARY OUTCOMES:
Sedentary behavior | one-week (168 hours) sit-and-stand desk cycle
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes standing/active during one week.
Sedentary behavior | one-week (168 hours) control cycle
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes per day standing/active.
Sedentary behavior | one-week (168 hours) cycloergometer cycle
  Sedentary behavior measured by actimetry using Actigraph® in number of minutes standing/active during one week.
Heart rate variability | 24 hours record corresponding to 12 hours of work and the next 12 hours of rest
  The heart rate variability measured using Zephyr®
Electrodermal activity | 24 hours record corresponding to 12 hours of work and the next 12 hours of rest
  The electrodermal activity measured using Empatica E4
Stress at home | 6 am, beginning of the control day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Stress at home | 6 am, beginning of the sit-and-stand desk day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Stress at home | 6 am, beginning of the cycloergometer day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Stress at home | 6 pm, end of the control day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Stress at home | 6 pm, end of the sit-and-stand desk day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Stress at home | 6 pm, end of the cycloergometer day
  Stress at home measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 am, beginning of the control day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 am, beginning of the sit-and-stand desk day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 am, beginning of the cycloergometer day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 pm, end of the control day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 pm, end of the sit-and-stand desk day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Fatigue | 6 pm, end of the cycloergometer day
  Fatigue measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 am, beginning of the control day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 am, beginning of the sit-and-stand desk day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 am, beginning of the cycloergometer day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 pm, end of the control day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 pm, end of the sit-and-stand desk day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Anxiety | 6 pm, end of the cycloergometer day
  Anxiety measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Mood | 6 pm, beginning of the control day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent). Higher scores mean a better outcome.
Mood | 6 am, beginning of the sit-and-stand desk day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent).Higher scores mean a better outcome.
Mood | 6 am, beginning of the cycloergometer day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent).Higher scores mean a better outcome.
Mood | 6 pm, end of the control day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent).Higher scores mean a better outcome.
Mood | 6 pm, end of the sit-and-stand desk day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent).Higher scores mean a better outcome.
Mood | 6 pm, end of the cycloergometer day
  Mood measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent).Higher scores mean a better outcome.
Stress at work | 6 am, beginning of the control day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Stress at work | 6 am, beginning of the sit-and-stand desk day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Stress at work | 6 am, beginning of the cycloergometer desk day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Stress at work | 6 pm, end of the control day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Stress at work | 6 pm, end of the sit-and-stand desk day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Stress at work | 6 pm, end of the cycloergometer day
  Stress at work measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum).Higher scores mean a worse outcome.
Amount of physical activity | 6 am, beginning of the control day
  Number of hours of physical activity during the last 24 hours
Intensity of physical activity | 6 am, beginning of the control day
  Physical activity intensity during the last 24 hours measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Amount of physical activity | 6 am, beginning of the sit-and-stand desk day
  Number of hours of physical activity during the last 24 hours
Intensity of physical activity | 6 am, beginning of the sit-and-stand desk day
  Physical activity intensity during the last 24 hours measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Amount of physical activity | 6 am, beginning of the cycloergometer day
  Number of hours of physical activity during the last 24 hours
Intensity of physical activity | 6 am, beginning of the cycloergometer day
  Physical activity intensity during the last 24 hours measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Amount of physical activity | 6 pm, end of the control day
  Number of hours of physical activity during the working day
Intensity of physical activity | 6 pm, end of the control day
  Physical activity intensity during the working day measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Amount of physical activity | 6 pm, end of the sit-and-stand desk day
  Number of hours of physical activity during the working day
Intensity of physical activity | 6 pm, end of the sit-and-stand desk day
  Physical activity intensity during the working day measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Amount of physical activity | 6 pm, end of the cycloergometer day
  Number of hours of physical activity during the working day
Intensity of physical activity | 6 pm, end of the cycloergometer day
  Physical activity intensity during the working day measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a higher intensity.
Sitting time | 6 am, beginning of the control day
  Number of hours sit during the last 24 hours
Sitting time | 6 am, beginning of the sit-and-stand desk day
  Number of hours sit during the last 24 hours
Sitting time | 6 am, beginning of the cycloergometer day
  Number of hours sit during the last 24 hours
Sitting time | 6 pm, end of the control day
  Number of hours sit during the working day
Sitting time | 6 pm, end of the sit-and-stand desk day
  Number of hours sit during the working day
Sitting time | 6 pm, end of the cycloergometer day
  Number of hours sit during the working day
Tabacco consumption | 6 am, beginning of the control day
  Number of cigarette during the last 24h
Tabacco consumption | 6 am, beginning of the sit-and-stand desk day
  Number of cigarette during the last 24h
Tabacco consumption | 6 am, beginning of the cycloergometer day
  Number of cigarette during the last 24h
Tabacco consumption | 6 pm, end of the control day
  Number of cigarette during the working day
Tabacco consumption | 6 pm, end of the sit-and-stand desk day
  Number of cigarette during the working day
Tabacco consumption | 6 pm, end of the cycloergometer day
  Number of cigarette during the working day
Tea consumption | 6 am, beginning of the control day
  Number of cups of tea during the last 24h
Tea consumption | 6 am, beginning of the sit-and-stand desk day
  Number of cups of tea during the last 24h
Tea consumption | 6 am, beginning of the cycloergometer day
  Number of cups of tea during the last 24h
Tea consumption | 6 pm, end of the control day
  Number of cups of tea during the last 24h
Tea consumption | 6 pm, end of the sit-and-stand desk day
  Number of cups of tea during the last 24h
Tea consumption | 6 pm, end of the cycloergometer day
  Number of cups of tea during the last 24h
Coffee consumption | 6 am, beginning of the control day
  Number of cups of coffee during the last 24h
Coffee consumption | 6 am, beginning of the sit-and-stand desk day
  Number of cups of coffee during the last 24h
Coffee consumption | 6 am, beginning of the cycloergometer day
  Number of cups of coffee during the last 24h
Coffee consumption | 6 pm, end of the control day
  Number of cups of coffee during the working day
Coffee consumption | 6 pm, end of the sit-and-stand desk day
  Number of cups of coffee during the working day
Coffee consumption | 6 pm, end of the cycloergometer day
  Number of cups of coffee during the working day
Sociodemographic | Once at baseline
  Sociodemographic will be assessed: gender, age, marital status, children, occupation, and recent stressful event
Sleep quality | Once at baseline
  Sleep quality measured using visual analogue scale ranging from 0 (Bad) to 100 (Excellent). Higher scores mean a better outcome.
Family support | Once at baseline
  Family support measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a better outcome.
Burnout | Once at baseline
  Burnout measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Job demand | Once at baseline
  Job demand measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a worse outcome.
Job control | Once at baseline
  Job control measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a better outcome.
Hierarchy support | Once at baseline
  Hierarchy support measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a better outcome.
Colleagues support | Once at baseline
  Colleagues support measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a better outcome.
Effort reward-imbalance | Once at baseline
  Effort reward-imbalance measured using visual analogue scale ranging from 0 (Minimum) to 100 (Maximum). Higher scores mean a better outcome.
Medical treatment | Once at baseline
  Medical treatment measured using multi-choice question "do you take long term medication?"
Allergy | Once at baseline
  Allergy measured using multi-choice question "do you have allergy?"
Average physical activity | Once at baseline
  Average number of hours of physical activity per week
Average physical activity intensity | Once at baseline
  Average physical activity intensity per week
Average tabacco consumption | Once at baseline
  Average number of cigarette per day
Average alcohol consumption | Once at baseline
  Average number of alcohol glasses per week
Average cannabis consumption | Once at baseline
  Average number of cannabis joint per week
Average tea consumption | Once at baseline
  Average number of cup of tea per day
Average coffee consumption | Once at baseline
  Average number of cup of coffee per day
Average food consumption | Once at baseline
  Average food consumption of 16 food groups
Diet characterization | Once at baseline
  "How do you characterize your diet" measured on a visual analogue scale ranging from 0 (Not at all balanced) to 100 (Very balanced)
RPAQ questionnaire | Once at baseline
  The Recent Physical Activity Questionnaire (RPAQ) assesses the level of physical activity and sedentary lifestyle in adults over the past four weeks. It is divided into three parts: work and study, home and leisure, and finally, stairs and travel. It makes it possible to classify individuals into several categories, one on sedentary lifestyle (low, resistant either 3-7h/day or high or >7h/day) and one on the level of physical activity (<8.3 Metabolic equivalent of task(MET).hour/week: inactive or >8.3 MET.h/wk: active).
MBI questionnaire | Once at baseline
  The Maslach Burn-out Inventory (MBI) is composed of 22 items designed to assess the three components of the burn-out syndrome: emotional exhaustion (9 items), depersonalization (5 items) and reduced personal accomplishment (8 items). The items are written in the form of statements about personal feelings or attitudes. Items are made of a 7-point scale frequency of feelings, varying from "never" to "every day". The scores for each component of the burn-out syndrome are considered separately. If desired for participant feedback, each score can be coded as low, average, or high.
JDCS questionnaire | Once at baseline
  The Job Demand-Control-Support (JDCS) questionnaire of Karasek assess job demands, job control and social support through 26 items. The questionnaire measures nine items of job demands, nine items of job control and eight items of social support. Items of JDCS are scored on a four-point Likert-type scale, ranging from 1 = strongly disagree to 4 = strongly agree. Among the 26 items, five negative statements require reverse scoring. From French data, the job strain threshold is set for a demands score higher than 20 and a control score lower than 71; the isostrain threshold is determined from a combining score of job strain and social support lower than 24. We would ask the participants to fulfil the questionnaire from memories that they keep of their work.
ERI questionnaire | Once at baseline
  The Effort-Reward Imbalance Questionnaire (ERI) is a self-administrated test assessing psychological distress and health problems that may occur when there is an imbalance between the efforts required by the work and the rewards received. We used the 46 items of the French version of the ERI model exploring efforts (six items), over commitment (eleven items), and rewards (seventeen items). Items of ERI were scored on a five-point Likert-type scale, ranging from 1 = disagree to 5 = agree and very disturbed. A ratio extrinsic efforts and rewards can assess the imbalance between these two dimensions. A ratio greater than one defines employees exposed to an imbalance between efforts and rewards.
Salivary cortisol | 6 am, beginning of the control day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 am, beginning of the control day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 am, beginning of the control day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 am, beginning of the control day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 9 am on the control day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 9 am on the control day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 9 am on the control day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 9 am on the control day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 12 am on the control day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 12 am on the control day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 12 am on the control day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 12 am on the control day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 3 pm on the control day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 3 pm on the control day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 3 pm on the control day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 3 pm on the control day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 6 pm, end of the control day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 pm, end of the control day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 pm, end of the control day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 pm, end of the control day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 6 am, beginning of the sit-and-stand desk day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 am, beginning of the sit-and-stand desk day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 am, beginning of the sit-and-stand desk day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 am, beginning of the sit-and-stand desk day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 9 am on the sit-and-stand desk day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 9 am on the sit-and-stand desk day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 9 am on the sit-and-stand desk day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 9 am on the sit-and-stand desk day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 12 am on the sit-and-stand desk day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 12 am on the sit-and-stand desk day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 12 am on the sit-and-stand desk day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 12 am on the sit-and-stand desk day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 3 pm on the sit-and-stand desk day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 3 pm on the sit-and-stand desk day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 3 pm on the sit-and-stand desk day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 3 pm on the sit-and-stand desk day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 6 pm, end of the sit-and-stand desk day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 pm, end of the sit-and-stand desk day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 pm, end of the sit-and-stand desk day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 pm, end of the sit-and-stand desk day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 6 am, beginning of the cycloergometer day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 am, beginning of the cycloergometer day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 am, beginning of the cycloergometer day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 am, beginning of the cycloergometer day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 9 am on the cycloergometer day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 9 am on the cycloergometer day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 9 am on the cycloergometer day
  Salivary leptin measured in ng/dml
Salivary ghrelin | 9 am on the cycloergometer day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 12 am on the cycloergometer day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 12 am on the cycloergometer day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 12 am on the cycloergometer day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 12 am on the cycloergometer day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 3 pm on the cycloergometer day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 3 pm on the cycloergometer day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 3 pm on the cycloergometer day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 3 pm on the cycloergometer day
  Salivary ghrelin measured in ng/ml
Salivary cortisol | 6 pm, end of the cycloergometer day
  Salivary cortisol measured in µg/dl
Salivary DHEAS | 6 pm, end of the cycloergometer day
  Salivary DHEAS measured in pg/ml
Salivary leptin | 6 pm, end of the cycloergometer day
  Salivary leptin measured in ng/ml
Salivary ghrelin | 6 pm, end of the cycloergometer day
  Salivary ghrelin measured in ng/ml
Blood cortisol | 6 am, beginning of the cycloergometer day
  Blood cortisol measured in ng/ml or nmol/l
Blood cortisol | 6 pm, end of the cycloergometer day
  Blood cortisol measured in ng/ml or nmol/l
Blood DHEAS | 6 am, beginning of the cycloergometer day
  Blood DHEAS measured in µg/ml
Blood DHEAS | 6 pm, end of the cycloergometer day
  Blood DHEAS measured in µg/ml
Blood leptin | 6 am, beginning of the cycloergometer day
  Blood leptin measured in ng/ml
Blood leptin | 6 pm, end of the cycloergometer day
  Blood leptin measured in ng/ml
Blood ghrelin | 6 am, beginning of the cycloergometer day
  Blood ghrelin measured in pg/ml
Blood ghrelin | 6 pm, end of the cycloergometer day
  Blood ghrelin measured in pg/ml
Blood BDNF | 6 am, beginning of the cycloergometer day
  Blood brain-derived neurotrophic factor (BDNF) measured in pg/ml
Blood BDNF | 6 pm, end of the cycloergometer day
  Blood brain-derived neurotrophic factor (BDNF) measured in pg/ml
Blood pro-inflammatory cytokines | 6 am, beginning of the cycloergometer day
  Blood pro-inflammatory cytokines measured in pg/ml
Blood pro-inflammatory cytokines | 6 pm, end of the cycloergometer day
  Blood pro-inflammatory cytokines measured in pg/ml
Blood NPY | 6 am, beginning of the cycloergometer day
  Blood vascular distribution of neuropeptide Y (NPY) measured in pg/ml
Blood NPY | 6 pm, end of the cycloergometer day
  Blood vascular distribution of neuropeptide Y (NPY) measured in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Fréderic DUTHEIL, Principal Investigator — fdutheil@chu-clermontferrand.fr
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes
After contacting the corresponding author and signing a data sharing agreement, investigators will make available the documents and personal data strictly necessary in accordance with laws and regulations (Articles L.1121-3 and R.5121-13 of the Code of Public Health).
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Clinchamps M, Bouillon-Minois JB, Trousselard M, Schmidt J, Pic D, Taillandier T, Mermillod M, Pereira B, Dutheil F. Effects of a sedentary behaviour intervention in emergency dispatch centre phone operators: a study protocol for the SECODIS randomised controlled cross-over trial. BMJ Open. 2024 Oct 9;14(10):e080177. doi: 10.1136/bmjopen-2023-080177. PMID 39384224